CLINICAL TRIAL: NCT02824744
Title: Comparison Between 2l/Min/kg vs 3l/Min/kg in High Flow Nasal Cannula (HFNC) During the Initial Management of Severe Bronchiolitis in Infants
Brief Title: Comparison Between 2l vs 3l in HFNC During the Initial Management of Severe Bronchiolitis in Infants
Acronym: TRAMONTANE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9719
Record Dates: First submitted 2016-06-27; First posted 2016-07-07 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2016-07

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; High flow nasal canula
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment by 2l/min/kg in HFNC (Active Comparator): treatment by 2l/min/kg in High Flow Nasal cannula (HFNC) during the initial management of severe bronchiolitis in infants (0-6 months years old)
  Interventions: Device: treatment by 2l/min/kg in High Flow Nasal cannula (HFNC)
- treatment by 3l/min/kg in HFNC (Experimental): treatment by 3l/min/kg in High Flow Nasal cannula (HFNC) during the initial management of severe bronchiolitis in infants (0-6 months years old)
  Interventions: Device: treatment by 3l/min/kg in High Flow Nasal cannula (HFNC)

INTERVENTIONS:
Device: treatment by 2l/min/kg in High Flow Nasal cannula (HFNC)
  Arms: treatment by 2l/min/kg in HFNC
Device: treatment by 3l/min/kg in High Flow Nasal cannula (HFNC)
  Arms: treatment by 3l/min/kg in HFNC

SUMMARY:
The purpose of the study is to evaluate prospectively the clinical benefits of 2 different flow with High flow nasal canula (HFNC: 2l/kg/min) versus (HFNC: 2l/kg/min) in the initial management of bronchiolitis in infants.

Design: Prospective, controlled, randomized, multi-center.

Design: Infants less than 6 month admitted in pediatric intensive care unit for respiratory distress (mWCAS >3) secondary to bronchiolitis but not requiring mechanical ventilation will be randomized in two groups:HFNC "2l/min/kg" or HFNC "3l/min/kg" during 24 hours.

Conditions of measurements:

Primary endpoint: Proportion of failure in both arms during the first 24 hours.

Failure criteria: A raise of the Clinical score for respiratory distress (mWCAS) (1 point) or respiratory rate (10/min /H0 and above 60/min) or discomfort (EDIN) (1point /H0 and above 4) or apnea.

Secondary outcomes: Assessment at H1, H12, H24 of mWCAS, respiratory and heart rate, EDIN score, skin lesions, FiO2 required to achieve an oxygen saturation between 94 and 97%, transcutaneous PCO2 (correlated to an initial gas analysis), Report SpO2 / FiO2

Statistic: Intention to treat Analysis.

Expected number of patients: 135 per arm: 270 children.

ELIGIBILITY:
Inclusion Criteria:

* age < 6 months
* bronchiolitis
* mWCAS > or =3
* hospitalisation: PICU
* signed consent form by parents

Exclusion Criteria:

* Intubated patient
* Neurological or cardiac disease

Ages: 0 Hours to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Proportion of failure in both arms | up to 24 hours
  Proportion of failure in both arms during the first 24 hours. Failure criteria: A raise of the Clinical score for respiratory distress (mWCAS) (1 point) or respiratory rate (10/min /H0 and above 60/min) or discomfort (EDIN) (1point /H0 and above 4) or apnea.

SECONDARY OUTCOMES:
assessment of heart rate in both arm | up to 24 hours
Assessment of the discomfort in both arms with the score of EDIN | up to 24 hours
assessment of the fraction of inspired oxygen (FiO2) in both arms | up to 24 hours
  FiO2 required to achieve an oxygen saturation between 94 and 97%
number of participants with an aggravation of the clinical score for respiratory distress arms (mWCAS) | up to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
All data will be centralized at the sponsor office for the final analysis

REFERENCES:
- [Derived] Milesi C, Pierre AF, Deho A, Pouyau R, Liet JM, Guillot C, Guilbert AS, Rambaud J, Millet A, Afanetti M, Guichoux J, Genuini M, Mansir T, Bergounioux J, Michel F, Marcoux MO, Baleine J, Durand S, Durand P, Dauger S, Javouhey E, Leteurtre S, Brissaud O, Renolleau S, Portefaix A, Douillard A, Cambonie G; GFRUP Respiratory Study Group. A multicenter randomized controlled trial of a 3-L/kg/min versus 2-L/kg/min high-flow nasal cannula flow rate in young infants with severe viral bronchiolitis (TRAMONTANE 2). Intensive Care Med. 2018 Nov;44(11):1870-1878. doi: 10.1007/s00134-018-5343-1. Epub 2018 Oct 21. PMID 30343318